CLINICAL TRIAL: NCT01981317
Title: Stepped Care Cognitive Behavioral Therapy for Pediatric Obsessive Compulsive Disorder
Acronym: SC-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Obsessive Compulsive Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOCDF2013
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2018-10

CONDITIONS: Obsessive Compulsive Disorder; Stepped Care Cognitive Behavioral Therapy
Keywords: Obsessive Compulsive Disorder; Cognitive Behavioral Therapy; Stepped Care CBT; Exposure and Response Prevention; Psychotherapy; Counseling
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Stepped Care CBT (Experimental): All participants in this arm receive Step One which includes 3-in-office sessions lasting 1 hour each over 6 weeks and 6 weekly phone calls lasting 15 minutes or less. The in-office sessions are devoted to psychoeducation, cognitive therapy, and hierarchy development. These sessions will include all procedures of the standard therapist-delivered CBT but will be parent-led, therapist guided; thus, the parent is delivering evidence-based strategies with clinician guidance.
  Children are then "stepped up" to Step Two of SC-CBT if it is determined that more therapy is needed following the post assessment. Step Two is a continuation of therapy and will include 9 additional in-office weekly session lasting 1 hour each over 9 weeks. These sessions will be therapist-led and are devoted to exposure and response prevention.
  Interventions: Behavioral: Stepped Care Cognitive Behavioral Therapy
- Standard CBT (Active Comparator): All patients in this arm will receive 12 sessions of therapy over 12 weeks using the evidence-based cognitive behavioral therapy protocol in POTS (2004). Sessions 1-3 do not include exposures and are devoted to psychoeducation, cognitive therapy, and hierarchy development. Sessions 4-12 involve exposure and response prevention exercises specific to each youth.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Stepped Care Cognitive Behavioral Therapy
  Arms: Stepped Care CBT
Behavioral: Cognitive Behavioral Therapy
  Arms: Standard CBT

SUMMARY:
The purpose of this research study is to determine how well children with OCD can be helped using therapy that requires less clinic visits. The investigators are testing a Stepped-Care Cognitive Behavioral Therapy (SC-CBT) approach in which children receive a full course of parent-led, therapist-guided treatment for OCD. The goal is to see if therapy can be done in fewer visits to the clinic. Children receiving SC-CBT will start with Step One, which includes three therapy sessions over six weeks. Those who do not get better in Step One will "STEP UP" to Step Two which involves coming in to meet with a therapist for the remaining sessions. Youth receiving SC-CBT will be compared to youth receiving standard CBT in the clinic through this study. It is expected that Stepped Care will be an acceptable, cost-effect, and feasible treatment with outcomes similar to standard CBT.

DETAILED DESCRIPTION:
Below is a summary of assessment and interventions as part of the study (separated by condition). Two thirds will receive SC-CBT, one-third standard CBT (determined at random following the initial phone screen).

A. Phone Screen (with parent)

B. Informed Consent and Initial Assessment

C. Randomization to either SC-CBT or Standard CBT

D. Treatment Phase (either 1 or 2 determined at random following 'C')

1. SC-CBT

   Children who are randomized into SC-CBT will receive Step One:
   * 3-in-office sessions - 1 hour each (over 6 weeks)
   * 6 weekly phone calls (15 minutes or less)
   * Post assessment (at the end of the 6 weeks)
   * 3-month follow up

   Children are "stepped up" to Step Two of SC-CBT if we determine more therapy is needed (following the post assessment). Step Two is a continuation of therapy and will include:
   * 9-in-office weekly sessions - 1 hour each (over 9 weeks)
   * Post assessment (after session 9)
   * 3-month follow up

   OR
2. Standard CBT

Children who are randomized into the standard CBT group will receive:

* 12-in-office weekly sessions - 1 hour each (over 12 weeks)
* Midpoint Assessment (after 6 weeks)
* Post assessment (at the end of the 12 weeks)
* 3-month follow up

ELIGIBILITY:
Inclusion Criteria:

* Outpatient youth with obsessive-compulsive disorder between the ages 8-17 years.
* A Children's Yale-Brown Obsessive-Compulsive Scale score ≥ 16
* Child has a Full Scale IQ ≥ 80 as assessed on the WASI
* English speaking

Exclusion Criteria:

* Past adequate CBT with E/RP trial
* Initiation of antidepressant medication within 12 weeks before study enrollment, or an antipsychotic/mood stabilizer medication 6 weeks before study enrollment, or a stimulant/anxiolytic or alpha 2 agonist 4 weeks before study enrollment
* Established Treatment changes: Any change in dose of an established psychotropic medication (e.g., antidepressants) within 8 weeks before study enrollment (4 weeks for antipsychotic, mood stabilizer, alpha 2 agonist; 2 weeks for stimulant/anxiolytic). Alternative medications must be stable for 4 weeks prior to baseline. Any medications must remain stable during treatment; downward adjustments due to side effects may be acceptable with PI approval.
* Active child suicidality assessed by all available information (e.g., KSADS-PL, CDI).
* DSM-IV conduct disorder, autism, mental retardation, bipolar, schizophrenia/schizoaffective disorders; or substance abuse in past 6 months; or co-primary eating disorder; using all available information.
* Another behavioral/emotional problem or psychiatric disorder is considered to be more problematic than OCD.
* Non-English speaking.
* WASI-IQ SS <80.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2017-03 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale | 12 weeks
  The Children's Yale-Brown Obsessive-Compulsive Scale is a psychometrically sound clinician-rated interview assessing OCD symptom severity.
Clinical Global Impression Improvement Scale | 12 weeks
  The CGI-I is a widely used 7-point clinician rating of clinical improvement.

SECONDARY OUTCOMES:
Clinical Global Impression Severity Scale | 12 weeks
  The CGI-S is a widely used 7-point clinician rating of clinical severity.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lewin, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- The Rothman Center for Pediatric Neuropsychiatry, St. Petersburg, Florida, United States